CLINICAL TRIAL: NCT06403384
Title: Effects of Vibration Therapy on Muscle Soreness and Athletic Performance in Wheelchair Basketball Players
Brief Title: Vibration Therapy in Wheelchair Basketball Players
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karabuk University (Other)
Responsible Party: Principal Investigator, MERT UYSAL, Lecturer, Karabuk University
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: KBU-FTR-MU-01
Record Dates: First submitted 2024-04-30; First posted 2024-05-07 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2024-05

CONDITIONS: Wheelchair Users; Athletic Performance; Disability; Disabled Persons
Keywords: Athlete; Disabled persons; Exercise; Pain; Proprioception; Upper extremity
MeSH Terms: conditions — Motor Activity; Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): no intervention was applied for the control group
- Vibration (Experimental): Vibration was applied for the vibration group
  Interventions: Device: Vibration

INTERVENTIONS:
Device: Vibration — Local vibration was applied
  Arms: Vibration

SUMMARY:
No study was found that investigated the effect of vibration therapy (VT) on recovery from exercise in WCB players. Therefore, the aim of the study was to investigate the effects of wearable local vibration device on muscle soreness and athletic performance during recovery from exercise in the elbow area in WCB players.

DETAILED DESCRIPTION:
Vibration therapy (VT) has been widely used to increase performance and rehabilitate injuries in athletes. Delayed onset muscle soreness (DOMS), caused by excessive overload after training and competitions, leads to loss of performance. The aim of this study was to investigate the effects of wearable local VT on muscle soreness and athletic performance in wheelchair basketball (WCB) players.

ELIGIBILITY:
Inclusion Criteria:

* Being a wheelchair basketball players

Exclusion Criteria:

* Having had an upper extremity operation within the last 6 months

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2022-08-01 (Actual)

PRIMARY OUTCOMES:
Muscle Soreness | pre-exercise (baseline), and 30 minutes and 24 hours post-exercise
  Muscle soreness was evaluated for both arms of the athletes with the "Numeric Pain Scale". This scale is horizontally scored between 0-10 (0 = no pain, 10 = unbearable pain).
Shooting percentage | pre-exercise (baseline), and 30 minutes and 24 hours post-exercise
  The participants were asked to shoot 10 free throws in total from the free throw line with the wheelchair after a warmup. The percentage of successful throws was accepted as the shooting percentage value of the athletes (number of successful throws x 100 / total number of throws).
20-meter sprint test | pre-exercise (baseline), and 30 minutes and 24 hours post-exercise
  For the test, a 20-meter track was created on the basketball court floor, and 2 meters were added to the distance and marked so that the athletes would not slow down on the last meters. The time to complete the 20-meter track with the ready and start command of the participants was recorded with a stopwatch.
Joint position sense | pre-exercise (baseline), and 30 minutes and 24 hours post-exercise
  Joint position sense was evaluated with the passive to active joint repositioning method using a digital inclinometer device. The participants sat with the elbow extended and eyes closed on their wheelchairs. The target angles were selected 30°, 60° and 90° of the elbow joint.
Range of motion | pre-exercise (baseline), and 30 minutes and 24 hours post-exercise
  Both elbow joint extension/flexion angles were measured with a universal goniometer (baseline) with the arm in anatomical position on the wheelchair.

CONTACTS AND LOCATIONS:
Overall Officials: Mert Uysal, Principal Investigator — Karabuk University
Locations (1):
- Karabuk U, Karabük, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No